CLINICAL TRIAL: NCT03015584
Title: Systems Biology Approach to Cognitive Impairment After SepsiS (CASS)
Brief Title: Systems Biology Approach to Cognitive Impairment After SepsiS
Acronym: CASS
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Samuel Brown, Director of Center for Humanizing Critical Care; Assistant Director of Critical Care Echocardiography Service, Intermountain Medical Center, Intermountain Health Care, Inc.
Other Study IDs: 1040524
Record Dates: First submitted 2016-12-08; First posted 2017-01-10 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Sepsis; Cognitive Impairment
MeSH Terms: conditions — Sepsis; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood for RNA-seq and whole exome sequencing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Septic patients admitted to the ICU

SUMMARY:
This study will use systems biology techniques, especially RNA-seq, to understand cognitive impairment after sepsis requiring an intensive care unit (ICU) admission.

ELIGIBILITY:
Inclusion Criteria

- Either SEPSIS or SEPTIC SHOCK

A. SEPSIS:

PRESENCE OF

1. Suspected or confirmed infection AND
2. Organ dysfunction as defined by a SOFA >= 2 above baseline (if no baseline data available, SOFA assumed to be 0)

OR

B. SEPTIC SHOCK:

AFTER INTRAVENOUS INFUSION OF 20ML/KG CRYSTALLOID OR EQUIVALENT, PRESENCE OF

1. Suspected or confirmed infection AND
2. Lactate > 2 mmol/L AND
3. Receiving vasopressors

Enrollment within 48 hours of ICU admission.

Must live within 200 miles of Intermountain Medical Center

Subject is at least 18 years of age or older

Must speak English

Exclusion Criteria:

* Onset of sepsis or septic shock >24 hours after hospital admission
* Patients transferred from another hospital except for directly from an emergency room
* Patients transferred to the ICU >48 hours after admission to Intermountain Medical Center (must have been admitted with diagnosis of sepsis)
* Prior traumatic brain injury, stroke, or intracranial hemorrhage
* DNR/DNI order before study enrollment
* Primary diagnosis of stroke or intracranial hemorrhage
* Known preexisting dementia or substantial cognitive impairment of any cause (established from both chart review, report and/or score ≥3 on IQ Code screening.
* Prior cardiac surgery (coronary artery bypass grafting or surgical valve replacement or repair)
* Known schizophrenia or other psychotic thought disorder
* Known pregnancy
* Primary diagnosis of drug overdose
* Attending physician deems aggressive care unsuitable
* Enrolled in another study if that study involves drug interventions
* Not expected to survive 48 hours
* Has a terminal condition independent of the acute illness that is expected to lead to death within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sepsis or septic shock, admitted to the ICU.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-06; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Hayling Sentence Completion test | 6 months
  Measures executive function. 6-month Hayling Sentence Completion test is the prespecified primary outcome.

SECONDARY OUTCOMES:
Wechsler Memory Scale Logical Memory 1 assessment | 3 months
Wechsler Memory Scale Logical Memory 1 assessment | 6 months
Wechsler Memory Scale Logical Memory 2 assessment | 3 months
Wechsler Memory Scale Logical Memory 2 assessment | 6 months
Digit Span memory assessment | 3 months
Digit Span memory assessment | 6 months
Verbal Fluency test | 3 months
Verbal Fluency test | 6 months
Wechsler Similarities assessment | 3 months
Wechsler Similarities assessment | 6 months
EuroQol five dimensions questionnaire (EQ-5D-3L) | 3 months
EuroQol five dimensions questionnaire (EQ-5D-3L) | 6 months
36-item short form survey (SF-36) | 3 months
36-item short form survey (SF-36) | 6 months
Hospital Anxiety and Depression Scale (HADS) | 3 months
Hospital Anxiety and Depression Scale (HADS) | 6 months
Impact of Event Scale-Revised (IES-R) | 3 months
Impact of Event Scale-Revised (IES-R) | 6 months
Functional Performance Inventory (FPI) | 3 months
Functional Performance Inventory (FPI) | 6 months
Functional Assessment of Chronic Illness Therapy (FACIT) | 3 months
Functional Assessment of Chronic Illness Therapy (FACIT) | 6 months
Activities of Daily Living/Instrumental Activities of Daily Living (ADL/IADL) | 3 months
Activities of Daily Living/Instrumental Activities of Daily Living (ADL/IADL) | 6 months
Hayling Sentence Completion test | 3 months

OTHER OUTCOMES:
90-day mortality | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Brown, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (1):
- Intermountain Medical Center, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown SM, Collingridge DS, Wilson EL, Beesley S, Bose S, Orme J, Jackson J, Hopkins RO. Preliminary Validation of the Montreal Cognitive Assessment Tool among Sepsis Survivors: A Prospective Pilot Study. Ann Am Thorac Soc. 2018 Sep;15(9):1108-1110. doi: 10.1513/AnnalsATS.201804-233OC. No abstract available. PMID 30168744